CLINICAL TRIAL: NCT06755671
Title: A Prospective Multicentre Real-world Assessment of the Efficacy of Danning Tablets in Alleviating Digestive Symptoms
Status: Recruiting | Type: Observational
Sponsor: Shanghai Hutchison Pharmaceuticals Limited (Industry)
Collaborators: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: CCPE202401
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2024-12

CONDITIONS: Indigestion; Dyspepsia; Bloating; Loss of Appetite; Reflux Acid; Constipation; Upper Abdominal Pain; Functional Dyspepsia
Keywords: Danning Tablets; dyspepsia; indigestion; observational study; real world study
MeSH Terms: conditions — Dyspepsia; Anorexia; Gastroesophageal Reflux; Constipation; Abdominal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with dyspepsia symptoms taking Danning Tablets: 1. Patients between 18 and 75 years old;
  2. Patients with at least one of the following symptoms: upper abdominal pain, bloating, loss of appetite, acid reflux or constipation;
  3. Patients already taking Danning Tablets as part of their regular medicine treatment for dyspepsia;
  4. Patients agree to sign the informed consent form.
  Interventions: Drug: Danning Tablet

INTERVENTIONS:
Drug: Danning Tablet — Danning Tablet is the only exposure in this observational study.

SUMMARY:
The goal of this observational study is to evaluate if Danning Tablets are effective in alleviating dyspepsia in patients with any of the following digestive symptoms: upper abdominal pain, bloating, loss of appetite, acid reflux or constipation.

The main questions it aims to answer are:

How effective are Danning Tablets for patients with indigestion symptoms? What are the impact factors (e.g. severity of conditions, demographic features, dose and length of treatment etc.) of the efficacy of Danning Tablets for indigestion patients?

Participants already taking Danning Tablets as part of their regular medical care for indigestion will take questionnaires by the end of two weeks and four weeks respectively from the start of their treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 75 years old
* Patients with at least one of the following symptoms: upper abdominal pain, bloating, loss of appetite, acid reflux or constipation
* Patients already taking Danning Tablets as part of their regular medicine treatment for dyspepsia
* Patients agree to sign the informed consent form

Exclusion Criteria:

* Past history or comorbidity of malignant tumor
* Comorbidity of severe systemic condition including cardiovascular, cerebrovascular, renal and hematopoietic system diseases
* Past history of abdominal surgery (post pancreatic surgery, post subtotal gastrectomy; incomplete intestinal obstruction) or mental illness, mobility difficulty (e.g. long-term bed ridden)
* Comorbidity of any unstable chronic or acute disease,which may impact the evaluation of treatment efficacy as determined by the research physician
* Pregnancy or breastfeeding
* Participation in other clinical trials within the past 3 months
* Other circumstances determined as ineligible by the research physician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with dyspepsia symptoms taking Danning Tablets
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Dyspepsia symptoms responder rate post treatment | From enrollment to the end of 4 weeks post enrollment
  A responder status is defined as patients reaching both a decrease of at least 50% regarding the Gastrointestinal Symptom Rating Scale (GSRS) score, and either symptom-free or markedly improved in the Global Patient Assessment (GPA) .
  GSRS consists of 15 items for assessment of gastrointestinal symptoms. The 15 items include five symptom clusters: Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation. Each item is rated on a 7-point Likert scale. The reliability and validity of the GSRS are well-documented. GSRS can be self-administered in approximately 3~5 minutes.
  The GPA asks patients the question "Please rate the strength of your upper abdominal complaints in the past 14 days. Please select how much they have changed compared to the condition at the onset of treatment: symptom-free, markedly improved, slightly improved, unchanged, worse".

SECONDARY OUTCOMES:
GPA responder rate | From enrollment to the end of 2 weeks and 4 weeks post enrollment
  A responder status is defined as patients reaching either symptom-free or markedly improved in the GPA.
GSRS score responder rate | From enrollment to the end of 2 weeks and 4 weeks post enrollment
  A responder status is defined as patients reaching a decrease of at least 50% regarding the GSRS score.
Abdominal pain rating | From enrollment to the end of 2 weeks and 4 weeks post enrollment
  Abdominal pain rating is defined as the multiplication of symptom frequency and severity rates. Abdominal pain frequency and severity are recorded in patient diary card. Symptom frequency is rated on a 5-point Likert scale. Symptom severity is rated through Visual Analogue Scale (VAS).
Quality of Life assessment through EQ-5D-5L | From enrollment to the end of 2 weeks and 4 weeks post enrollment
  TheEuroQol 5 Dimension 5-level (EQ-5D-5L) is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Adverse event rate | From enrollment to the end of 2 weeks and 4 weeks post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Jianting CAI, Doctor of Medicine, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The investigators have decided not to share IPD for confidentiality purpose. Yet IPD may be shared upon reasonable request on a one to one basis.